CLINICAL TRIAL: NCT01570842
Title: The Role of Anthropometry in Gastroesophageal Reflux Disease and Esophageal Injury
Brief Title: Anthropometry in Gastroesophageal Reflux Disease and Esophageal Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-005468
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal reflux disease; GERD; Barrett's esophagus
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anthropometric Measurements; Tissue Samples (Other): All participants will have their waist circumference and waist to hip ratio taken as a measurement of central obesity. Participants undergoing clinically indicated upper endoscopy and who consent to providing tissue samples will have 8 tissue samples taken for future research purposes.
  Interventions: Other: Anthropometric measurements; Procedure: Tissue samples

INTERVENTIONS:
Other: Anthropometric measurements — All participants will have their waist circumference and waist to hip ratio taken as a measurement of central obesity.
Procedure: Tissue samples — Participants undergoing clinically indicated upper endoscopy and who consent to providing tissue samples will have 8 tissue samples taken for future research purposes.

SUMMARY:
Is waist to hip ratio (WHR), waist circumference (WC), (as markers of visceral adiposity) associated with an increase in acidic and non acidic reflux as well as systemic inflammation involving esophageal mucosa, thereby increasing esophageal injury and predisposing to subsequent development of Barrett's esophagus (BE)?

DETAILED DESCRIPTION:
The investigators will study 100 adult subjects over the age of 18 from the esophageal motility lab who are undergoing clinically indicated 24 hour acidity or basicity (pH) impedance and/or pH studies off acid suppressing medication.. These subjects will not have a prior history of esophageal surgery, or diagnosis of BE. The investigators will obtain consent for taking anthropometric measurements (Waist and hip circumference), and the results of their study. Only those subjects that successfully complete the 24 hour pH impedance studies will be included. Subjects will also undergo clinically indicated endoscopy. The investigators will consent these subjects to obtain 4 biopsies (bx) from the gastroesophageal (GE) junction and 4 bx from 5 cm above the GE junction. These bio-specimens will be stored for assessment of tissue injury (PGE2) and tissue immune-histochemistry of BE precursors (CDX1 and CDX2) at a later date.

ELIGIBILITY:
Inclusion:

* Subjects over the age of 18 undergoing clinically indicated 24 hour pH impedance and/or pH studies. Many will also undergo clinically indicated endoscopy, and consent for acquiring tissue samples for future biomarker staining tests will be obtained.
* Able to give informed consent

Exclusion:

* Subjects with a prior history of esophageal surgery, or diagnosis of BE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Correlate Anthropometry with number of acid reflux episodes | 1 year
  To correlate measures of central obesity waist/hip ratio (WHR) and waist circumference (WC) with number of reflux episodes (acidic and non acidic), and other measures of acid/non acid reflux. Stratify by use of proton pump inhibitors (PPIs).

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States